CLINICAL TRIAL: NCT06238258
Title: Healthcare Outcomes of a Staff/Caregiver Training Program Focused on Challenging Behaivors for Adults With Developmental Disability and Co-occurring Mental Health Disorders
Brief Title: Dual Diagnosis Training Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, John Philips, Professor Emeritus, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-124
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Training Group
Keywords: intellectual disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Arm (Experimental)
  Interventions: Behavioral: SPECTROM Training

INTERVENTIONS:
Behavioral: SPECTROM Training — Training regarding treatment of behavioral challenges in adults with intellectual disability

SUMMARY:
This is a clinical trial, with participants undergoing the 16 hour SPECTROM training, and completing 2 assessments before and after training (the Psychotropic Knowledge Questionnaire-Revised and the Management of Aggression and Violence Attitude Scale-Revised-ID).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are individuals who work in the 3 ARCA group homes or in the UNM psychiatric center and who are fluent in English and 18 years and older

Exclusion Criteria:

* All participants must be fluent in English because for this pilot study we do not have funds to translate study materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Knowledge Acquisition Post Training | 6 months
  Completion of assessments

CONTACTS AND LOCATIONS:
Locations (1):
- UNM Health Science Center, Albuquerque, New Mexico, United States